CLINICAL TRIAL: NCT06469177
Title: Patient Centered Post-operative Pain Management Software Tool Vs Standard of Care: a Controlled Clinical Trial in Elective Shoulder, Hip and Knee Arthroplasty Patients.
Brief Title: Patient Centered Post-Op Pain Management Software Tool Interventional Study Verses Standard of Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64876
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Post-operative Pain, Acute; Opioid Use, Unspecified; Arthroplasty Complications; Knee Osteoarthritis; Shoulder Arthritis; Hip Arthritis
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized, parallel group prospective interventional study. Patient participants will be consented and then randomized to either the "treatment group" and a "control group".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Coach App Users (Experimental): Participants enrolled in Pain Coach App software and directed to download on their mobile device
  Interventions: Device: Pain Coach App
- Standard of Care (No Intervention): Participants received traditional standard of care supports for joint arthroplasty surgery

INTERVENTIONS:
Device: Pain Coach App — Pain Coach App is a mobile application that offers patients undergoing shoulder, hip and knee arthroplasty surgery preoperative educational tools and questionnaires to provide patient specific details to their surgeons for prescribing purposes as well as post operative pain assessment and medication reminders/tracking, problem troubleshooting and a resource library for further pain management tools and education.
  Arms: Pain Coach App Users

SUMMARY:
The goal of this clinical trial is to learn if the Pain Coach App will result in less opioids being prescribed to and used by patients undergoing Shoulder/Hip/Knee Arthroplasty surgery while maintaining the same or better pain control versus standard of care. The main questions it aims to answer are:

1. Will elective shoulder, hip and knee arthroplasty patients using PainCoach App be prescribed and/or use less opioids, measured by total morphine milliequivalents (MME) after surgery when compared to those treated as standard of care while maintaining similar pain control?
2. Will arthroplasty surgeons using PainCoach App write more patient-specific prescriptions resulting in a reduction in opioids prescribed after surgery with no increase in further opioids prescribed in the months following surgery?
3. Will the use of Pain Coach App lead to equal or reduced healthcare system utilization after surgery?
4. Will patients and surgeons using PainCoach App find it helpful enough to use it again and recommend to colleagues, family and friends?

Researchers will compare participants assigned to use Pain Coach App vs participants assigned to standard of care arm to see if there are differences in opioid prescriptions and self reported use.

Participants will either use the Pain Coach App or follow standard of care instructions and be followed forward for the opioid prescriptions dispensed in community and self-reported opioids use at study end.

DETAILED DESCRIPTION:
This will be a randomized, parallel group prospective interventional study. Patient participants will be consented and then randomized using a tool built into RedCap to either the "treatment group" and a "control group". The treatment group will be sent an email with instructions to set up a Pain Coach Account and download the app onto their mobile device. (Phone or tablet)The control group will not be offered Pain Coach technology and will just follow the usual care pathway for arthroplasty patients. When a participant in the treatment arm completes the initial questionnaire within the app (known as the Pain Coach Profile) this information will be used by a pharmacist in the study to create a suggested prescription for that patient. This suggested prescription will be provided to the patients surgeon for them to review and either accept, edit or discard based on their own clinical judgement.- For the rest of the study the patients in the treatment arm will have access to the Pain Coach app functionalities and use them as they require/prefer. A survey will be sent to both treatment and control groups after their surgery on Post Op Day 2 and 30 to assess pain control. There will be an interim analysis once 281 participants have been recruited into each treatment arm. At this point a retrospective chart review will be used to identify ED related visits for surgical pain within 90 days will be compared between groups at 6 months, also the amount of opioids prescribed (and number of refills) up to 3 months after surgery will be recorded and compared between groups. If at this point there is a statistically significant difference between groups the study will end early. Otherwise it will control until 561 participants are assigned to each group. This will provide 80% power to detect a minimally clinically important difference of 10% reduction in opioid prescribing between groups.

ELIGIBILITY:
Inclusion Criteria:

* Elective total shoulder (day surgery only), hip or knee arthroplasty completed within NSH, starting at the HI or DGH
* OR date for surgery is known and booked
* Able to access the internet via mobile device (has access to smart phone)
* If expresses concern about low tech IQ, has a support person available
* Able to read and write in English

Exclusion Criteria:

* Non-elective arthroplasty surgery procedures (trauma, fractures)
* Bilateral knee or hip arthroplasty
* Unable to read or write in English
* Lacks capacity to provide consent due to cognitive impairment
* No access to internet or mobile device to use self-help pain management tools
* Inpatient Shoulder arthroplasty as residents write these discharge prescriptions

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Opioid Prescriptions Efficacy Information | At discharge, 2 weeks, 1 and 3 months after surgery.
  Describe and compare immediate release opioids prescription quantities (in MME) filled by patients and surgeons using PainCoach App vs Standard of Care.
Pain Related Adverse Effects | Post Operative Day 2 and 30
  Assess for any Pain/Opioid related side effects by administering the QoR-15 questionnaire (see appendix to both groups and reviewing ED visits by patients in both treatment and control groups to ensure safety/efficacy of application use.

SECONDARY OUTCOMES:
Health Systems Usage | From discharge to 90 days post-op
  Describe patient reported interactions with the healthcare system including patient reported calls to surgeon's office, calls to the Orthopedic Assessment Clinic, calls to their primary care provider and calls to their pharmacy as a composite endpoint
Self reported Opioid usage | At Post Op Day 30
  Describe and compare patients' self-reported usage of opioids after surgery.
  1. How many days after surgery did they use opioids?
  2. Did the patient use all of the opioids they were prescribed? (Yes/no)
  i. If no: How many opioid tablets did have left after surgery will be used to compare to amount originally filled to report absolute MME used after surgery for each treatment group.
Surgeon Adoption | Study End
  Describe satisfaction and compliance with PainCoach App prescribing tools.
  1. Were surgeons satisfied with the prescriptions and progress notes provided by PainCoach App?
  2. Frequency surgeon followed one of three pathways: if they used the full suggested prescription, made changes or used their default prescribing pathway ? Which will be identified via chart review.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health QEII and Dartmouth General Hospital, Dartmouth, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pain Coach Inc. Website — http://www.paincoachapp.com